CLINICAL TRIAL: NCT03239704
Title: Improving Outcomes Among Urgent Care Clinic Patients With Inflammatory Bowel Disease (URGENT-IBD)
Brief Title: Improving Outcomes Among Urgent Care Clinic Patients With Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Crohn's and Colitis Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: URGENT-IBD
Record Dates: First submitted 2017-08-02; First posted 2017-08-04 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Inflammatory Bowel Disease; Ulcerative Colitis; Crohn Disease
Keywords: Inflammatory Bowel Disease; Ulcerative Colitis; Crohn Disease; Quality Improvement; Telemedicine
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Follow-Up and Telemedicine Monitoring (Experimental)
  Interventions: Behavioral: Telemedicine Follow-Up; Other: Telemedicine Monitoring; Behavioral: 30 Day Comprehensive Questionnaire
- Minimal Intervention (Active Comparator)
  Interventions: Behavioral: 30 Day Comprehensive Questionnaire

INTERVENTIONS:
Behavioral: Telemedicine Follow-Up — Organized follow-up with an IBD advanced practice nurse at 24-48 hours, 7 days, and 30 days post-urgent care clinic appointment; to monitor the health status of patients with respect to their IBD.
  Arms: Telemedicine Follow-Up and Telemedicine Monitoring
Other: Telemedicine Monitoring — Patients will be provided access to a smartphone application entitled: 'Health Promise'. The application will generate short questionnaires every 3 days, where patients can self-report their Crohn's disease activity as measured by the PRO-2 score or Ulcerative Colitis activity as measured by the 6-Point Mayo score, and medication adherence as measured by the MMAS-8 scale. The survey responses will be monitored by an IBD advanced practice nurse, to arrange for additional telemedicine follow-up sessions or to triage patients for an expedited appointment with a gastroenterologist.
  Arms: Telemedicine Follow-Up and Telemedicine Monitoring
Behavioral: 30 Day Comprehensive Questionnaire — Patients will complete a web-based questionnaire at 30 days following the urgent care clinic visit when they were enrolled in the study. The questionnaire will query the following: Patient Demographics; Patient Satisfaction as measured by the CACHE Questionnaire; IBD related Quality of Life as measured by the IBDQ questionnaire; and Crohn's Disease activity as measured by the PRO-2 score or Ulcerative Colitis Activity as measured by the 6-Point Mayo score.

SUMMARY:
Inflammatory Bowel Diseases (IBD) refers to a category of disorders, consisting of Crohn's Disease (CD) and Ulcerative Colitis (UC), where segments of the gastrointestinal tract become inflamed and ulcerated. Canada has among the highest incidence rates of IBD in the world - 16.3 and 12.3 per 100,000 for CD and UC respectively. In the absence of a cure, the current goal of treatment is to manage patients in a milder state of remission. However, maintaining (or even achieving) remission is dependent on timely access to specialist IBD care; which in light of rising incidence rates have proven to be challenging. Moreover, patients often experience flare-ups of their gastrointestinal symptoms, while awaiting access to specialist care. In recent years, there has been increased integration of telemedicine services in gastroenterology practice. This change has been driven by a desire among IBD patients to have more flexible follow-up care, where 'virtual' care is provided as an adjunct to in-person consultations. Within the context of IBD, telemedicine might be effective in delivering routine and timely follow-up care to high-risk patients. The purpose of this study to determine whether telemedicine-based follow-up care can effectively manage the gastrointestinal symptoms of high-risk IBD patients and reduce their need for preventive health care services.

DETAILED DESCRIPTION:
Inflammatory Bowel Diseases (IBD) refers to a category of disorders, consisting of Crohn's Disease (CD) and Ulcerative Colitis (UC), where segments of the gastrointestinal tract become inflamed and ulcerated. Canada has among the highest incidence rates of IBD in the world - 16.3 and 12.3 per 100,000 for CD and UC respectively. Moreover, IBD care spans a broad range of inpatient, outpatient, and emergency services; which vary across populations due to the heterogeneous nature of these conditions. The economic burden of IBD in Canada is estimated to be $2.8 billion per anum, where direct health care costs (i.e. medications, hospitalizations, physician visits) alone exceed $1.2 billion.

In the absence of a cure, the current goal of treatment is to manage patients in a milder state of remission. However, maintaining (or even achieving) remission is dependent on timely access to specialist IBD care; which in light of rising incidence rates have proven to be challenging. Wait times for gastroenterology care are currently in excess of guidelines outlined by the Canadian Association of Gastroenterology - Wait Times Consensus Group. Moreover, patients often experience flare-ups of their gastrointestinal symptoms, while awaiting access to specialist care.

In recent years, there has been increased integration of telemedicine services in gastroenterology practice. This change has been driven by a desire among IBD patients to have more flexible follow-up care, where 'virtual' care is provided as an adjunct to in-person consultations. Telemedicine is the process by which medical information is transferred between providers and patients through an electronic interface (i.e. two-way video, smartphone applications and secure messaging). Within the context of IBD, telemedicine might be effective in delivering routine and timely follow-up care to high-risk patients. It's also enticing to speculate that if telemedicine follow-up care can adequately manage the gastrointestinal symptoms of high-risk patients, then it may also reduce their need for preventive health care services and alleviate some of the economic burden associated with these conditions.

Therefore, the purpose of this study to determine whether telemedicine-based follow-up care can effectively manage the gastrointestinal symptoms of high-risk IBD patients and reduce their need for preventive health care services. As part of this study, we will attempt to recruit all IBD outpatients, who were seen at the Mount Sinai Hospital urgent care clinic. These are a subset of high-risk IBD patients, who often have moderate to severe exacerbations of their medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Confirmed diagnosis of Crohn's Disease or Ulcerative Colitis
* Recruited from an IBD urgent care clinic

Exclusion Criteria:

* Subjects who can't communicate in English
* Subjects who are read or write in English
* Subjects who lack internet access
* Subjects who lack access to a personal smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Post-Appointment IBD related Hospital Admission | Within 30 days of study enrolment
  Incidence of post-appointment IBD related hospital admission will be recorded for all patients enrolled in the study. Post-appointment hospital admissions will be defined as any IBD related hospital admission following the initial urgent care clinic appointment when the patient was enrolled in the study. Post-appointment IBD related hospital admission rates will will be compared between study groups.

SECONDARY OUTCOMES:
Post-Appointment IBD related Surgery | Within 30 days of study enrolment
  Incidence of post-appointment IBD related surgery will be recorded for all patients enrolled in the study. Post-appointment IBD related surgery will be defined as any IBD related surgery following the initial urgent care clinic appointment when the patient was enrolled in the study. Post-appointment IBD related surgery rates will be compared between compared study groups
Patient Satisfaction with Health Care in IBD | At 30 days following study enrolment
  Patient satisfaction with health care in IBD as measured by CACHE will be collected from all patients, through a web-based questionnaire administered at 30 days following the initial urgent care clinic appointment, where the patient was enrolled in the study. Mean scores for Patient Satisfaction with Health Care in IBD will be compared between study groups.
IBD related Quality of Life | At 30 days following study enrolment
  IBD related Quality of Life as measured by IBDQ will be collected from all patients, through a web-based questionnaire administered at 30 days following the initial urgent care clinic appointment, where the patient was enrolled in the study. Mean scores for IBD related Quality of Life will be be compared between study groups.
Disease Activity | At 30 days following study enrolment
  Disease Activity as measured by PRO-2 score for Crohn's Disease or the 6-Point Mayo score for Ulcerative Colitis will be collected from all patients, through a web-based questionnaire administered at 30 days following the initial urgent care clinic appointment where the patient was enrolled in the study. Mean scores for disease activity will be compared between study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey C Nguyen, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rocchi A, Benchimol EI, Bernstein CN, Bitton A, Feagan B, Panaccione R, Glasgow KW, Fernandes A, Ghosh S. Inflammatory bowel disease: a Canadian burden of illness review. Can J Gastroenterol. 2012 Nov;26(11):811-7. doi: 10.1155/2012/984575. PMID 23166905
- [Background] Park MD, Bhattacharya J, Park K. Differences in healthcare expenditures for inflammatory bowel disease by insurance status, income, and clinical care setting. PeerJ. 2014 Sep 23;2:e587. doi: 10.7717/peerj.587. eCollection 2014. PMID 25279267
- [Background] Novak K, Veldhuyzen Van Zanten S, Pendharkar SR. Improving access in gastroenterology: the single point of entry model for referrals. Can J Gastroenterol. 2013 Nov;27(11):633-5. doi: 10.1155/2013/519342. Epub 2013 Sep 13. PMID 24040629
- [Background] Paterson WG, Depew WT, Pare P, Petrunia D, Switzer C, Veldhuyzen van Zanten SJ, Daniels S; Canadian Association of Gastroenterology Wait Time Consensus Group. Canadian consensus on medically acceptable wait times for digestive health care. Can J Gastroenterol. 2006 Jun;20(6):411-23. doi: 10.1155/2006/343686. PMID 16779459
- [Background] Paterson WG, Barkun AN, Hopman WM, Leddin DJ, Pare P, Petrunia DM, Sewitch MJ, Switzer C, van Zanten SV. Wait times for gastroenterology consultation in Canada: the patients' perspective. Can J Gastroenterol. 2010 Jan;24(1):28-32. doi: 10.1155/2010/912970. PMID 20186353
- [Background] Cross RK, Kane S. Integration of Telemedicine Into Clinical Gastroenterology and Hepatology Practice. Clin Gastroenterol Hepatol. 2017 Feb;15(2):175-181. doi: 10.1016/j.cgh.2016.09.011. Epub 2016 Dec 16. No abstract available. PMID 27989663
- [Background] Kemp K, Griffiths J, Campbell S, Lovell K. An exploration of the follow-up up needs of patients with inflammatory bowel disease. J Crohns Colitis. 2013 Oct;7(9):e386-95. doi: 10.1016/j.crohns.2013.03.001. Epub 2013 Mar 27. PMID 23541150